CLINICAL TRIAL: NCT04854083
Title: Semaglutide as an Adjunct to Dieting in the Treatment of Type 2 Diabetes - Effects on Glucose Metabolism, Prevention of Weight Regain and Peripheral Tissue Metabolic Activation
Brief Title: Semaglutide as an Adjunct to Dieting in the Treatment of Type 2 Diabetes
Acronym: MitoSema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kirsi Pietiläinen (Other)
Collaborators: University of Helsinki (Other); Turku University Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Kirsi Pietiläinen, Professor, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Type2 Diabetes
Keywords: weight loss; dieting
MeSH Terms: conditions — Weight Loss | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): The intervention study for the patients with T2DM begins with a low-calorie diet (LCD) phase run-in for 13 weeks. During re-introduction of food, the participants will be assigned to semaglutide 1.34mg/ml treatment for 44 weeks (dose escalation in total 8 weeks, maintenance period for 36 weeks).
  Interventions: Drug: Semaglutide, 1.34 mg/mL
- Placebo (Placebo Comparator): The intervention study for the patients with T2DM begins with a low-calorie diet (LCD) phase run-in for 13 weeks. During re-introduction of food, the participants will be assigned to placebo treatment for 44 weeks (dose escalation in total 8 weeks, maintenance period for 36 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide, 1.34 mg/mL — The low-calorie diet (LCD) has a phase run-in period for 13 weeks for all participants including 8 weeks of total LCD followed 5-week gradual re-introduction of food (replacement of the VLCD products by one meal/week). During re-introduction of food, the subjects will be randomly assigned to semaglutide 1.34mg/ml (subcutaneous administration, dose escalation 0.25 mg once weekly for 4 weeks, 0.5 mg once weekly for 4 weeks, where after 1.0 mg once weekly) until the end of the study (12 months). The participants will receive lifestyle counselling throughout the study.
  Other Names: Ozempic
  Arms: Semaglutide
Drug: Placebo — The low-calorie diet (LCD) has a phase run-in period for 13 weeks for all participants including 8 weeks of total LCD followed 5-week gradual re-introduction of food (replacement of the VLCD products by one meal/week). During re-introduction of food, the subjects will be randomly assigned to placebo (subcutaneous administration, dose escalation 0.25 mg once weekly for 4 weeks, 0.5 mg once weekly for 4 weeks, where after 1.0 mg once weekly) until the end of the study (12 months). The participants will receive lifestyle counselling throughout the study.
  Arms: Placebo

SUMMARY:
The pharmacological approaches in the treatment of type 2 diabetes (T2DM) have advanced radically during the last decades. However, focus on long-term management of body weight, which is an essential part of treatment success, is often lacking. Excluding surgery, there are only a few effective treatment methods for obesity. Management of obesity is also greatly challenged by weight regain, which is common after a successful lifestyle intervention. Weight regain typically results in the deterioration of glucose homeostasis in T2DM. However, understanding the pathomechanisms of weight regain and subsequent worsening of glucose homeostasis is still insufficient. Therefore, T2DM treatment programs that target long-term weight management have been scarce. This study aims to fill the gaps in the current knowledge by advancing the development of treatment programs for T2DM that simultaneously head for improved glucose metabolism and improved long-term body weight control.

DETAILED DESCRIPTION:
In this randomized, double-blind, parallel, placebo-controlled trial we compare the effects of semaglutide 1.34 mg/ml vs. normal dieting by randomizing the patients with both T2DM and overweight/obesity (BMI ≥27) (n=50, aged ≥18 to < 65 years) to two groups: both groups participate in a similar lifestyle treatment to induce weight loss, but one group gets an add-on of semaglutide 1.34mg/ml while the other is treated with placebo. Additionally, a reference group of healthy normal weight non-diabetic individuals (BMI ≤ 25 kg/m2, n=25, aged ≥18 to < 65 years) are included as controls at the initiation of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and <65 years
* BMI: ≥27 kg/m2
* T2DM (HbA1c ≥ 6.0% if on anti-diabetic medication or HbA1c≥6.5% if non- medicated)
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Contraindication to trial drugs
* Use of insulin or GLP-1RAs (during the past 3 months)
* Use of anti-obesity drugs (during the past 3 months)
* Weight change of >5% during the past 3 months
* Bariatric surgery or planned bariatric surgery during the trial
* History of pancreatitis
* Impaired renal function (GFR<30 ml/min/1.73m2)
* Impaired hepatic function (ALAT>2 x upper limit normal)
* Clinically significant active cardiovascular disease
* Clinically significant abnormality in the ECG
* Cancer (except basal or squamous cell skin cancers)
* Major psychiatric disease (such as severe depression, bipolar disorder, schizophrenia)
* Substance abuse
* Learning disability
* Females of childbearing potential not using adequate contraceptive methods
* Pregnancy
* Lactation
* Any other condition that in the opinion of the investigator could interfere with the conduction of the study or interpretation of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
HbA1c | from baseline to 12 months
  Change in HbA1c (%)

SECONDARY OUTCOMES:
HbA1c | from baseline to 6 months
  Change in HbA1c (%)
Fasting plasma glucose | from baseline to 6 and 12 months
  Change in fasting plasma glucose (mmol/l)
Body weight | from baseline to 6 and 12 months
  Change in body weight (kg)
Percentage of patients reaching ≥5%,10% & 15% weight loss | from baseline to 6 and 12 months
Waist circumference | from baseline to 6 and 12 months
  Change in waist circumference (cm)
Change in appetite and eating habits, control of eating | from baseline to 6 and 12 months
  Using questionnaire Control of Eating (CoEQ)
Change in appetite and eating habits, binge eating | from baseline to 6 and 12 months
  Using questionnaires Binge Eating Scale(BES), Questionnaire on Eating and Weight Patterns (QEWP)
Change in appetite and eating habits, emotional, external and restraint eating | from baseline to 6 and 12 months
  Using questionnaire Dutch Eating Behaviour Questionnaire (DEBQ)
Blood pressure | from baseline to 6 and 12 months
  Change in blood pressure (mmHg)
Plasma lipids | from baseline to 6 and 12 months
  Change in lipids (total cholesterol, LDL, HDL, TAG) (mmol/l)
Changes in concomitant antidiabetic medications | from baseline to 6 and 12 months
  Change in number of antidiabetic medications
Changes in concomitant antihypertensive medications | from baseline to 6 and 12 months
  Change in number of antihypertensive medications
Changes in concomitant lipid medications | from baseline to 6 and 12 months
  Change in number of lipid medications
Mitochondrial DNA quantification | from baseline to 6 and 12 months
  Change in mitochondrial DNA (mtDNA) copy number, RNA expression of mtDNA encoded genes in adipose tissue and skeletal muscle
Change in the transcriptomics profile of adipose tissue and skeletal muscle | from baseline to 6 and 12 months
  Change in the transcriptomics profile by qPCR and/or RNA sequencing
Change in the oxygen uptake and perfusion in subcutaneous and intra-abdominal adipose tissue, brown adipose tissue, skeletal muscle, gut and liver | from baseline to 12 months
  Change in the oxygen uptake and perfusion measured by PET/CT (in vivo)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Pietiläinen, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- University of Helsinki, Helsinki, Finland